CLINICAL TRIAL: NCT01161069
Title: A Double Blind (3rd Party Open), Randomized, Placebo Controlled, Parallel Group, Multiple Dose Escalation Study To Evaluate The Safety, Toleration, Pharmacokinetics Of PF-03049423 In Healthy Young Adult Volunteers And Healthy Elderly Volunteers
Brief Title: A Study To Evaluate The Safety And Tolerability Of Different Doses Of PF-03049423 In Healthy Adult Volunteers And Healthy Older Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A9541002
Record Dates: First submitted 2010-05-07; First posted 2010-07-13 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: phase 1; healthy young adult volunteers; healthy elderly adult volunteers
MeSH Terms: interventions — 3-(4-(2-hydroxyethyl)piperazin-1-yl)-7-(6-methoxypyridin-3-yl)-1-(2-propoxyethyl)pyrido(3,4-b)pyrazin-2(1H)-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-03049423 (Active Comparator): Cohorts 1 through 3 were healthy young adult volunteers; cohorts 4 and 5 were healthy elderly adult volunteers
  Interventions: Drug: PF-03049423
- Drug (Placebo Comparator): Placebo in oral solution, given once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-03049423 — PF-03049423 in oral solution, 2.5 mg, given once daily for 14 days; healthy young adult volunteers
  Arms: PF-03049423
Drug: PF-03049423 — PF-03049423 in oral solution, 7.5 mg, given once daily for 14 days; healthy young adult volunteers
  Arms: PF-03049423
Drug: PF-03049423 — PF-03049423 in oral solution, 6 mg, given once daily for 7 days, then 12 mg given once daily for 7 days; healthy young adult volunteers
  Arms: PF-03049423
Drug: PF-03049423 — PF-03049423 in oral solution, 3 mg, given once daily for 7 days, then 6 mg given once daily for 7 days; healthy elderly adult volunteers
  Arms: PF-03049423
Drug: PF-03049423 — PF-03049423 in oral solution, 5 mg, given once daily for 7 days, then 10 mg given once daily for 7 days; healthy elderly adult volunteers
  Arms: PF-03049423
Drug: Placebo — Placebo in oral solution, given once daily for 14 days
  Arms: Drug

SUMMARY:
The purpose this study is to evaluate the safety and toleration of PF-03049423 following multiple dose administration as an oral solution to healthy young adult volunteers and healthy elderly volunteers. The study will also evaluate the pharmacokinetics of PF-03049423 after multiple dose administration to healthy young adult volunteers and healthy elderly volunteers. The study will also explore the relationship between blood pressure (supine and standing) and PF-03049423 concentration.

DETAILED DESCRIPTION:
The purpose of the investigation is to evaluate the safety and tolerability of an investigational new drug, PF-03049423, when dosed for two weeks in both healthy younger and healthy older subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons, male or female.
* For the healthy young adult cohort, subjects must be 18 to 50 years old, inclusive.
* For the healthy elderly adult cohort, subjects must be 51 to 99 years old, inclusive.
* Body Mass Index (BMI) of 18 to 35; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Subjects with clinically significant medical conditions.
* Women of non-child bearing potential.
* Subjects with a known medical history of hearing loss/disability or nonarteritic ischemic optic neuropathy.
* A positive urine drug screen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety laboratory assessments, vital signs (including supine and standing blood pressure), physical examination, 12-lead ECGs and adverse events. | Days 1 through 14
PK Parameters:Day 1: Area under concentration time curve from hour 0 to the last dosing interval (AUCtau), maximum observed concentration (Cmax), and time of maximum observed concentration (Tmax), for PF-03049423 in plasma. | Day 1
PK Parameters: Day 14: Cmax at steady state, Tmax, AUCtau at steady state , t½, Cavg at steady state, Cmin at steady state, Cmax at steady state /Cmax sd, AUCtau at steady state/ AUCtau sd, Ae% and CLr. | Day 14

SECONDARY OUTCOMES:
Blood pressure | Days 1 to 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9541002&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20Different%20Doses%20Of%20PF-03049423%20In%20Healthy%20Adult%20Volunteers%20And%20Healthy%20Older%20Volunt